CLINICAL TRIAL: NCT05631340
Title: The Effects Of Discharge Education Program On Recovery And Quality Of Life After Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Eva Kajti, Lecturer, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Eva Kajti
Record Dates: First submitted 2022-11-21; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Cardiac Surgery, Heart Surgery, Discharge Education, Nursing, Telenursing, m-Health, Quality of Life, Recovery
Keywords: Cardiac Surgery, Heart Surgery, Discharge Education, Nursing, Telenursing, m-Health, Quality of Life, Recovery

STUDY DESIGN:
Intervention Model Description: same follow up time
Who Masked: Participant
Masking Description: participants do not know the group they belong, case or control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- case group (Experimental): Recieving additional discharge education by the researcher and supported by a booklet and mobile app
  Interventions: Other: Discharge education
- control group (Active Comparator): Recieving standart hoapital discharge education
  Interventions: Other: Discharge education

INTERVENTIONS:
Other: Discharge education — Researcher's newly prepared discharge education supported by a booklet and mobile app

SUMMARY:
This study aims to build a new discharge education, booklet and mobile application based, and assess it's efffects on recovery and quality of life in cardiac surgery patients. This is a randomised control trial. 12 weeks follow up will be done by phone calls.

DETAILED DESCRIPTION:
Patients following cardiac surgery will be part of the study. Patients will be randomized in control and case groups. Control group receive standart discharge eduation from the nurses of the hospital, they will be interviewed by the researcher to gather general information and also information about recovery and quality of life. Case group will be given a discharge education by the researcher before discharge. After education patients will be given a booklet and a mobile application with the neccasary discharge information. Both groups will be followed for 12 weeks by monthly phone calls. In the last call recovery and quality of life will be reassesed.

ELIGIBILITY:
Inclusion Criteria:

* To agree to participate in the research,
* Open heart surgery patients
* Being 18 years or older,
* Being able to read, write, understand and communicate in Turkish,
* No vision, hearing and perception problems,
* Being conscious, oriented, cooperative and open to communication.

Exclusion Criteria:

• Having surgery other than open heart surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Recovery status after cardiac surgery | 12 weeks
  Recovery -40 Questionnaire mesure recovery status before discharge and 12 weeks after discharge
Quality of Life after cardiac surgery | 12 weeks
  Multidimensional Index of Life Quality questionnaire to mesure QoL before discharge and 12 weeks after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Ayfer Özbaş, Study Chair — Istanbul University-Cerrahpasa Florence Nightingale Faculty of Nursing
Locations (1):
- Istanbul Univesity-Cerrahpasa Florence Nightingale Faculty of Nursing, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Research data will be given statistically without sharing IPD